CLINICAL TRIAL: NCT00717613
Title: Psychosocial and Patient Education Needs of Prostate Cancer Patients Selecting Watchful Waiting
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, David Latini, Adjunct Assistant Professor of Urology, Baylor College of Medicine
Other Study IDs: DLD2007-01; NCT00729066 (obsolete NCT alias)
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Localized Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Observational cohort study

SUMMARY:
This study includes an interview with men who have selected "watchful waiting" or "active surveillance" for their localized prostate cancer, in lieu of active treatment (such as surgery or radiation). We hope to understand the educational and support needs of men on surveillance so that we can develop a new intervention that will improve quality of life for such men.

DETAILED DESCRIPTION:
Interviews are conducted over the telephone and require approximately 90 minutes to complete. Men interviewed are compensated for their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* 1) male,
* 2) 18 years or older, with biopsy-proven prostate cancer,
* 3) diagnosed with localized disease within the last 24 months,
* 4) have a telephone at the time of enrollment,
* 5) have an address where they can receive study materials by mail (a street address or post office box),
* 6) able to speak and understand English;
* 7) have selected surveillance, rather than active treatment for his prostate cancer.

Exclusion Criteria:

* 1) female
* 2) no diagnosis of localized prostate cancer
* 3) completed or undergoing active treatment (e.g., surgery, radiotherapy, etc.)
* 4) no phone or US mail address
* 5) unwilling or unable to provide informed consent
* 6) unable to speak and understand English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sample of men on active surveillance drawn from large academic medical centers, community hospitals, support groups, and the internet.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life, particularly cancer-specific anxiety and general anxiety | One time retrospective interview

CONTACTS AND LOCATIONS:
Overall Officials: David M Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States